CLINICAL TRIAL: NCT04683029
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, Proof-of-concept Study of Guselkumab in Participants With Systemic Sclerosis
Brief Title: A Study of Guselkumab in Participants With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108936; CNTO1959SSC2001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Guselkumab (Experimental): Participants will receive intravenous (IV) injection of Guselkumab Dose 1 at Week 0, 4, and 8 followed by subcutaneous (SC) injection of Dose 2 Guselkumab every 4 weeks (Q4W) from Week 12 to Week 48 (end of maintenance phase). Participants will receive SC injection of Guselkumab Dose 2 and IV injection of placebo at long-term extension (LTE) Weeks 52, 56, and 60 followed by SC injection of Guselkumab Dose 2 Q4W from LTE Week 64 until Week 100.
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 2
- Group B: Placebo (Placebo Comparator): Participants will receive IV injection of matching placebo at Week 0, 4, and 8 followed by SC injection of matching placebo Q4W from Week 12 to Week 48 (end of maintenance phase). Participants will receive SC injection of Placebo and IV injection of Guselkumab Dose 1 at LTE Weeks 52, 56, and 60 followed by SC injection of Guselkumab Dose 2 Q4W from LTE Week 64 until Week 100.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab Dose 1 — Guselkumab Dose 1 will be administered intravenously.
  Arms: Group A: Guselkumab
Drug: Guselkumab Dose 2 — Guselkumab Dose 2 will be administered subcutaneously.
  Arms: Group A: Guselkumab
Drug: Placebo — Placebo will be administered intravenously or subcutaneously.
  Arms: Group B: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of guselkumab in participants with systemic sclerosis (SSc).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of systemic sclerosis (SSc) according to American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) 2013 criteria
* Diffuse cutaneous SSc according to the LeRoy criteria that is, skin fibrosis proximal to the elbows and knees in addition to acral fibrosis
* Disease duration of ≤36 months (defined as time from first non-Raynaud phenomenon manifestation).
* Greater than or equal to (>=) 10 and less than or equal to (<=) 22 modified Rodnan skin score (mRSS) units at screening and Week 0
* Forced vital capacity (FVC) >= 60 percent (%) of predicted at screening
* Diffusing capacity of the lung for carbon monoxide (DLCO) >= 40% of predicted (hemoglobin-corrected) at screening.
* Participants who meet 1 of the following criteria at screening: increase of >=3 mRSS units, compared with an assessment performed within the previous 2 to 6 months; Involvement of 1 new body area with an increase of >=2 mRSS units compared with an assessment performed within the previous 2 to 6 months; and Involvement of 2 new body areas with increase of >=1 mRSS units compared with the assessment within the previous 2 to 6 months

Exclusion Criteria:

* History of liver or renal insufficiency (estimated creatinine clearance below 60 milliliter per minute [mL/min]); significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has any known severe or uncontrolled SSc complications including hemoptysis, pulmonary hemorrhage, renal crisis
* Has an interstitial lung disease requiring oxygen therapy
* Has any rheumatic disease other than SSc such as rheumatoid arthritis (RA), polymyalgia rheumatica (PMR), systemic lupus erythematosus, polymyositis/dermatomyositis that could interfere with assessment of SSc
* Has a current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances. (or, in the investigator's opinion, any other concomitant medical condition that places the participant at risk by participating in this study)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (4):
- Japan (4):
  - Chukyo Hospital, Aichi
  - The University of Tokyo Hospital, Tokyo
  - Wakayama Medical University Hospital, Wakayama
  - University of Fukui Hospital, Yoshida

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with systemic sclerosis as per American College of Rheumatology and European League Against Rheumatism 2013 criteria with disease duration of less than or equal to (<=) 36 months and Modified Rodnan Skin Score ranged from greater than or equal to (>=) 10 to less than or equal to (<=) 22 units were randomized into the study.
Groups:
- Main Study: Group A: Guselkumab: Participants received guselkumab 400 milligrams (mg) intravenous (IV) infusion (induction dosing) at Weeks 0, 4, and 8 followed by guselkumab 200 mg subcutaneous (SC) injection (maintenance dosing) every 4 weeks (Q4W) from Week 12 until Week 48. After Week 52, participants who did not enter LTE underwent the safety follow up until Week 60.
- Main Study: Group B: Placebo: Participants received placebo (matched to guselkumab 400 mg) IV infusion (induction dosing) at Weeks 0, 4, and 8 followed by placebo (matched to guselkumab 200 mg) SC injection (maintenance dosing) Q4W from Week 12 until Week 48. After Week 52, participants who did not enter LTE underwent the safety follow up until Week 60.
- LTE Period: Group A: Guselkumab Then Guselkumab: Participants who received guselkumab and completed the main study (Week 0 through 52, that is, after the Week 48 evaluation, prior to Week 52 evaluation) and who, in the opinion of the investigator benefited from continued treatment, entered LTE period and received guselkumab 200 mg SC injection and placebo IV infusion at Weeks 52, 56, and 60 followed by guselkumab 200 mg SC injection q4w from Week 64 until Week 100. After Week 100, participants were followed up until Week 112.
- LTE Period: Group B: Placebo Then Guselkumab: Participants who received placebo and completed the main study (Week 0 through 52, that is, after the Week 48 evaluation, prior to Week 52 evaluation) and who, in the opinion of the investigator benefited from continued treatment, entered LTE period and received guselkumab 400 mg IV infusion and placebo SC injection at Weeks 52, 56, and 60 followed by guselkumab 200 mg SC injection q4w from Week 64 until Week 100. After Week 100, participants were followed up until Week 112.
Period: Main Study: Week 0-Week 60
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
Started | 29 | 27 | 0 | 0
Completed | 28 | 27 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Long-term Extension(LTE):Week52-Week 112
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
Started | 0 | 0 | 25 (Participants who completed the main study (Week 0 through 52) and who signed the informed consent form (ICF) before or at Week 52, to participate in the LTE.) | 26 (Participants who completed the main study (Week 0 through 52) and who signed the informed consent form (ICF) before or at Week 52, to participate in the LTE.)
Completed | 0 | 0 | 24 | 24
Not Completed | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (13.26) | 50.8 (12.18) | 51.1 (12.64)
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 years | 25 | 23 | 48
  65 years and over | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 47
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 27 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Change From Baseline in Modified Rodnan Skin Score (mRSS) at Week 24
Description: Change from baseline in mRSS at Week 24 was reported. The mRSS is an accepted clinical measure of skin thickness. The investigator assessed the thickening of the skin using the mRSS through simple palpation on 17 different skin sites in the fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (no thickening) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome.
Time Frame: Baseline and Week 24
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Score on a scale | -9.5 (0.74) | 3.1 (0.77)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Test type: Superiority; p < 0.001, MMRM model; LS Mean Difference = -12.6, 80% CI 2-sided [-13.8 to -11.4]

2. Secondary Outcome: Main Study: Change From Baseline in Modified Rodnan Skin Score at Week 52
Description: Change from baseline in mRSS at Week 52 was reported. The mRSS is an accepted clinical measure of skin thickness. The investigator assessed the thickening of the skin using the mRSS through simple palpation on 17 different skin sites in the fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (no thickening) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome.
Time Frame: Baseline and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Score on a scale | -9.3 (0.89) | 2.7 (0.93)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Test type: Superiority; LS Mean Difference = -12.0, 80% CI 2-sided [-13.3 to -10.7]

3. Secondary Outcome: Main Study: Percentage of Participants Who Experienced Worsening of Modified Rodnan Skin Score at Week 24 and Week 52
Description: The percentage of participants who experienced worsening of mRSS at Week 24 and Week 52 was reported. The worsening of mRSS was defined as an increase from baseline greater than or equal to (>=) 5 points and >=20 percent (%) in mRSS. The mRSS is an accepted clinical measure of skin thickness. The investigator assessed the thickening of the skin using the mRSS through simple palpation on 17 different skin sites in the fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (no thickening) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome.
Time Frame: Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Percentage of participants
  Week 24 | 3.4 | 25.9
  Week 52 | 20.7 | 77.8
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; Odds Ratio (OR) = 0.1, 80% CI 2-sided [0.0 to 0.3]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; Odds Ratio (OR) = 0.1, 80% CI 2-sided [0.0 to 0.2]

4. Secondary Outcome: Main Study: Percentage of Participants Who Achieved a Score of 0.6 in American College of Rheumatology Combined Response Index in Diffuse Cutaneous Systemic Sclerosis (ACR CRISS) at Week 24 and Week 52
Description: ACR CRISS is a composite endpoint. Firstly, participants were evaluated on not-improved criterion: new onset of renal crisis, >=15% decline in forced vital capacity [FVC] percent predicted relative to baseline, new onset of pulmonary arterial hypertension, and new onset of left ventricular failure. If yes, these participants were assigned probability score of 0.0. For remaining participants, percentage was based on CRISS domains: mRSS, FVC percent predicted, physician's global assessment, patient's global assessment and Health Assessment Questionnaire Disability-Index (HAQ-DI). Algorithm determines predicted probability of improvement from baseline by incorporating change in mRSS, FVC percent predicted, physician and patient global assessments and HAQ-DI. Outcome was a continuous variable between 0.0 and 1.0 (0 to 100%). Higher score=greater probability of improvement. ACR CRISS score >=0.60 was considered improved, while predicted probability below 0.60 was considered not improved.
Time Frame: Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Percentage of participants
  Week 24 | 86.2 | 3.7
  Week 52 | 79.3 | 3.7
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; Odds Ratio (OR) = 203.2, 80% CI 2-sided [42.1 to 980.6]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; Odds Ratio (OR) = 130.3, 80% CI 2-sided [28.2 to 601.9]

5. Secondary Outcome: Main Study: Change From Baseline in Forced Vital Capacity (FVC) at Week 24 and Week 52
Description: FVC was the total amount of air (in liters) exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying interstitial lung disease.
Time Frame: Baseline, Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Liters
  Week 24 | -51.9 (33.91) | -4.7 (35.78)
  Week 52 | -26.5 (30.42) | -12.3 (32.15)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; LS Mean Difference = -47.2, 80% CI 2-sided [-96.8 to 2.4]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; LS Mean difference = -14.2, 80% CI 2-sided [-57.2 to 28.8]

6. Secondary Outcome: Main Study: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 24 and Week 52
Description: Change from baseline in the percent predicted FVC at Week 24 and Week 52 was reported. FVC was the total amount of air (in liters) exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying interstitial lung disease.
Time Frame: Baseline, Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Percent predicted FVC
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Percent predicted FVC
  Week 24 | -0.7 (1.21) | -0.7 (1.26)
  Week 52 | -0.2 (1.17) | -0.4 (1.22)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; LS Mean Difference = -0.0, 80% CI 2-sided [-1.7 to 1.6]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; LS Mean Difference = 0.1, 80% CI 2-sided [-1.4 to 1.7]

7. Secondary Outcome: Main Study: Change From Baseline in the Measured Absolute Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) at Week 24 and Week 52
Description: DLCO is a measurement of the ability of the lungs to transfer gases from the air to the blood. DLCO is measured using the single breath method. Participants breathe in (inhale) air containing a very small, harmless amount of a tracer gas, such as carbon monoxide. Participants hold their breath for 10 seconds, then rapidly blow it out (exhale). The exhaled gas was tested to determine amount of the tracer gas absorbed during the breath.
Time Frame: Baseline, Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Milliliter/minute/millimeter mercury
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Milliliter/minute/millimeter mercury
  Week 24 | -0.60 (0.257) | -0.51 (0.265)
  Week 52 | -0.35 (0.316) | -0.56 (0.327)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; LS Mean Difference = -0.08, 80% CI 2-sided [-0.44 to 0.27]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; LS Mean Difference = 0.21, 80% CI 2-sided [-0.29 to 0.71]

8. Secondary Outcome: Main Study: Change From Baseline in the Percent Predicted Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) at Week 24 and Week 52
Description: Change from baseline in the percent predicted DLCO at Week 24 and Week 52 was reported. DLCO is a measurement of the ability of the lungs to transfer gases from the air to the blood. DLCO is measured using the single breath method. Participants breathe in (inhale) air containing a very small, harmless amount of a tracer gas, such as carbon monoxide. Participants hold their breath for 10 seconds, then rapidly blow it out (exhale). The exhaled gas was tested to determine amount of the tracer gas absorbed during the breath.
Time Frame: Baseline, Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Percent predicted DLCO
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Percent predicted DLCO
  Week 24 | -4.57 (1.338) | -2.49 (1.347)
  Week 52 | -1.71 (1.541) | -1.85 (1.565)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; LS Mean Difference = -2.08, 80% CI 2-sided [-3.81 to -0.34]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; LS Mean Difference = 0.14, 80% CI 2-sided [-2.13 to 2.42]

9. Secondary Outcome: Main Study: Change From Baseline in Digital Ulcer Counts at Week 24 and Week 52
Description: Digital ulcers were defined as a full thickness (>3 millimeters [mm] in maximal diameter) skin lesion with loss of epithelium including lesions covered by eschar (excluding pitting scars and hyperkeratotic lesions). Healing was defined by re-epithelialization with loss of pain and exudate. The digital ulcer assessments and counting were performed by the investigator designee.
Time Frame: Baseline, Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Ulcers
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Ulcers
  Week 24 | -0.0 (0.47) | 4.8 (0.48)
  Week 52 | -0.1 (0.55) | 4.1 (0.58)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; LS Mean Difference = -4.9, 80% CI 2-sided [-5.7 to -4.0]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; LS Mean Difference = -4.3, 80% CI 2-sided [-5.1 to -3.5]

10. Secondary Outcome: Main Study: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24 and Week 52
Description: HAQ-DI assessed the degree of difficulty participants experienced in 8 daily living activity domains during past week: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each activity category consisted of 2-3 items. For each item, level of difficulty was scored from 0 to 3 (0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do). Total HAQ-DI score was computed as the sum of domain scores divided by the number of domains answered, providing a score from 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability.
Time Frame: Baseline, Week 24 and Week 52
Population: The FAS included all randomized participants who received at least 1 dose (complete or partial) of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Score on a scale
  Week 24 | -0.0529 (0.09062) | 0.3477 (0.09439)
  Week 52 | -0.0572 (0.08955) | 0.1782 (0.09321)
Statistical Analysis 1: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 24; Test type: Superiority; LS Mean Difference = -0.4006, 80% CI 2-sided [-0.5344 to -0.2668]
Statistical Analysis 2: Comparison: Main Study: Group A: Guselkumab vs Main Study: Group B: Placebo; Week 52; Test type: Superiority; LS Mean Difference = -0.2355, 80% CI 2-sided [-0.3730 to -0.0980]

11. Secondary Outcome: Main Study: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Through Week 24 and Week 52
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were defined as AEs that occur at or after the initial administration of study intervention. All TEAEs including serious and non-serious events are reported in this outcome measure.
Time Frame: From Baseline (Week 0) up to Week 24 and Week 52
Population: The safety analysis set included all randomized participants who received at least 1 dose (complete or partial) of study intervention. Participants were analyzed based on the intervention they received, regardless of the intervention groups to which they were assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Participants
  Week 24 | 20 | 24
  Week 52 | 25 | 26

12. Secondary Outcome: Long-term Extension (LTE) Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were defined as AEs that occurred at or after the initial administration of study intervention. All TEAEs including serious and non-serious events are reported in this outcome measure.
Time Frame: From Week 52 up to Week 112
Population: The safety analysis set for LTE period included all randomized participants who received at least 1 dose (complete or partial) of study intervention during LTE period.
Measure: Count of Participants; unit: Participants
Arm/Group | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
Number analyzed (Participants) | 25 | 26
Participants | 23 | 25

13. Secondary Outcome: Main Study: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) Through Week 24 and Week 52
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/ incapacity, or resulted in congenital anomaly/birth defect. TEAEs were defined as AEs that occur at or after the initial administration of study intervention.
Time Frame: From Baseline (Week 0) up to Week 24 and Week 52
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Participants
  Week 24 | 0 | 0
  Week 52 | 1 | 1

14. Secondary Outcome: Long-term Extension (LTE) Period: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: as for outcome 13
Time Frame: From Week 52 up to Week 112
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
Number analyzed (Participants) | 25 | 26
Participants | 1 | 0

15. Secondary Outcome: Main Study: Number of Participants With Adverse Events of Special Interest (AESI) Through Week 24 and Week 52
Description: AESI were defined as any newly identified malignancy or case of active tuberculosis (TB) or interstitial lung disease (ILD) occurring after the first study intervention administration in study participants and was reported by the investigator to the sponsor or designee within 24 hours after being made aware of the event. AESIs for this study included drug-induced liver injuries, active TB, ILD, hypersensitivity reaction, opportunistic infection and adverse cardiovascular events.
Time Frame: From Baseline (Week 0) up to Week 24 and Week 52
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo
Number analyzed (Participants) | 29 | 27
Participants
  Week 24 | 0 | 0
  Week 52 | 1 | 2

16. Secondary Outcome: Long-term Extension (LTE) Period: Number of Participants With Adverse Events of Special Interest (AESI)
Description: as for outcome 15
Time Frame: From Week 52 up to Week 112
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
Number analyzed (Participants) | 25 | 26
Participants | 0 | 0

17. Secondary Outcome: Main Study: Serum Concentration of Guselkumab
Description: Serum concentration of guselkumab was reported. The lower limit of quantification (LLOQ) for guselkumab was 0.01 micrograms per milliliter (mcg/mL).
Time Frame: Pre-dose at Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and Post- dose at Weeks 0, 4, 8
Population: Pharmacokinetics analysis set included all participants who received at least 1 complete administration of guselkumab and had at least 1 observed post dose PK data. Here, 'n' (number analyzed) refers to participants evaluable at specified time points. This outcome measure was planned to be analyzed for specified arm only.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Main Study: Group A: Guselkumab
Number analyzed (Participants) | 29
mcg/mL
  Pre-dose at Week 0 | NA (NA) — Since concentration was below LLOQ, hence mean and standard deviation could not be calculated.
  Post-dose at Week 0: number analyzed (Participants) | 28
  Post-dose at Week 0 | 140.880 (26.5879)
  Pre-dose at Week 4 | 22.489 (6.9499)
  Post-dose at Week 4 | 160.691 (31.7578)
  Pre-dose at Week 8 | 27.968 (9.7988)
  Post-dose at Week 8 | 164.633 (28.9999)
  Pre-dose at Week 12 | 36.497 (13.7929)
  Pre-dose at Week 16 | 21.697 (9.6355)
  Pre-dose at Week 20: number analyzed (Participants) | 28
  Pre-dose at Week 20 | 12.751 (6.0638)
  Pre-dose at Week 24 | 13.981 (6.6055)
  Pre-dose at Week 28: number analyzed (Participants) | 27
  Pre-dose at Week 28 | 14.184 (5.6980)
  Pre-dose at Week 32: number analyzed (Participants) | 26
  Pre-dose at Week 32 | 12.564 (5.6367)
  Pre-dose at Week 36: number analyzed (Participants) | 25
  Pre-dose at Week 36 | 12.932 (6.4345)
  Pre-dose at Week 40: number analyzed (Participants) | 25
  Pre-dose at Week 40 | 13.375 (6.1989)
  Pre-dose at Week 44: number analyzed (Participants) | 25
  Pre-dose at Week 44 | 12.469 (6.8698)
  Pre-dose at Week 48: number analyzed (Participants) | 25
  Pre-dose at Week 48 | 12.074 (6.1027)
  Pre-dose at Week 52: number analyzed (Participants) | 25
  Pre-dose at Week 52 | 11.363 (6.6822)

18. Secondary Outcome: Long-term Extension (LTE) Study: Serum Concentrations of Guselkumab
Description: Serum concentration of guselkumab was reported. The LLOQ for guselkumab was 0.01 mcg/mL.
Time Frame: Pre-dose (at Weeks 56, 60, 64, 76, 88, 96) and Week 104
Population: Pharmacokinetics analysis set included all participants who received at least 1 complete administration of guselkumab and had at least 1 observed post dose PK data. Here, 'n' (number analyzed) refers to participants analyzed at specified time points.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
Number analyzed (Participants) | 25 | 26
mcg/mL
  Pre-dose at Week 56 | 12.167 (5.4753) | 19.285 (8.3377)
  Pre-dose at Week 60 | 12.704 (5.6942) | 25.925 (10.9856)
  Pre-dose at Week 64 | 13.835 (7.3326) | 33.368 (14.8075)
  Pre-dose at Week 76: number analyzed (Participants) | 24 | 24
  Pre-dose at Week 76 | 11.641 (5.5746) | 13.200 (6.0810)
  Pre-dose at Week 88: number analyzed (Participants) | 24 | 24
  Pre-dose at Week 88 | 10.339 (5.1209) | 11.893 (6.3203)
  Pre-dose at Week 96: number analyzed (Participants) | 24 | 24
  Pre-dose at Week 96 | 10.082 (4.5371) | 12.426 (5.6925)
  Week 104: number analyzed (Participants) | 23 | 24
  Week 104 | 10.080 (5.2596) | 12.301 (6.0099)

19. Secondary Outcome: Main Study: Number of Participants With Anti-Guselkumab Antibody
Description: Number of participants with anti-guselkumab antibody were reported. Serum samples were assessed for anti-drug antibodies.
Time Frame: From Baseline (Week 0) up to Week 52
Population: Immunogenicity analysis set included all participants who received at least 1 administration of guselkumab and had at least 1 observed post dose immune response data. This outcome measure was planned to be analyzed for specified arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Group A: Guselkumab
Number analyzed (Participants) | 29
Participants | 6

20. Secondary Outcome: Long-term Extension (LTE) Study: Number of Participants With Anti-guselkumab Antibody
Description: as for outcome 19
Time Frame: From Week 52 up to Week 104
Population: Immunogenicity analysis set included all participants who received at least 1 administration of guselkumab and had at least 1 observed post dose immune response data.
Measure: Count of Participants; unit: Participants
Arm/Group | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
Number analyzed (Participants) | 25 | 26
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: Main Study: From screening (Week [-6]) up to Week 60 and LTE Period: From Week 52 up to Week 112 ; SAEs and Non-serious AEs: Main Study: From baseline (Week 0) up to Week 60; LTE Period: From Week 52 up to Week 112
Description: The safety analysis set included all randomized participants who received at least 1 dose (complete or partial) of study intervention during main study and LTE period. During LTE, AEs were analyzed per treatment group as participants received guselkumab and placebo at the same time so AEs per intervention could not be determined.
Arm/Group | Main Study: Group A: Guselkumab | Main Study: Group B: Placebo | LTE Period: Group A: Guselkumab Then Guselkumab | LTE Period: Group B: Placebo Then Guselkumab
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27 | 1/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/27 | 1/25 | 0/26
Other Adverse Events (participants affected / at risk) | 22/29 | 26/27 | 22/25 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Group A: Guselkumab (N=29) | Main Study: Group B: Placebo (N=27) | LTE Period: Group A: Guselkumab Then Guselkumab (N=25) | LTE Period: Group B: Placebo Then Guselkumab (N=26)
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Group A: Guselkumab (N=29) | Main Study: Group B: Placebo (N=27) | LTE Period: Group A: Guselkumab Then Guselkumab (N=25) | LTE Period: Group B: Placebo Then Guselkumab (N=26)
Tinnitus (Ear and labyrinth disorders) | 0 | 3 | 0 | 1
Conjunctival Haemorrhage (Eye disorders) | 1 | 0 | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Malaise (General disorders) | 3 | 3 | 0 | 0
Pyrexia (General disorders) | 9 | 14 | 4 | 7
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 0
Covid-19 (Infections and infestations) | 2 | 2 | 7 | 6
Cystitis (Infections and infestations) | 1 | 2 | 1 | 2
Dermatophytosis of Nail (Infections and infestations) | 0 | 2 | 0 | 0
Folliculitis (Infections and infestations) | 3 | 3 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Herpes Zoster (Infections and infestations) | 1 | 1 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 6 | 2 | 12 | 9
Paronychia (Infections and infestations) | 4 | 5 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 1
Streptococcal Infection (Infections and infestations) | 0 | 0 | 2 | 0
Tinea Pedis (Infections and infestations) | 2 | 3 | 0 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 3 | 3 | 3 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 3
Lymphocyte Count Decreased (Investigations) | 0 | 3 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 7 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 2 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 7 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 5 | 4 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 7 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04683029/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT04683029/SAP_001.pdf